CLINICAL TRIAL: NCT02794649
Title: Descriptive Analysis of Gut Microbiome Alterations in Hyperoxaluric Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: VA New York Harbor Healthcare System (U.S. Federal Agency)
Collaborators: Mayo Clinic (Other); New York University (Other)
Responsible Party: Principal Investigator, Lama Nazzal, MD, MSc, VA New York Harbor Healthcare System
Other Study IDs: RKSC6416
Record Dates: First submitted 2016-05-25; First posted 2016-06-09 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Oxalate, Primary Hyperoxaluria, Microbiome
MeSH Terms: conditions — Hyperoxaluria, Primary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — fecal samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- healthy: Individuals without a history of kidney or bowel disease
- primary hyperoxaluria: Patients diagnosed with type I PH by genetic testing
- enteric hyperoxaluria: Patients with Roux-en-Y-gastric-bypass.
- calcium oxalate stone formers: History of passing or having surgically removed a calcium oxalate kidney stone within 5 years of recruitment.

SUMMARY:
To characterize the microbiome in 4 groups of subjects (primary hyperoxaluria type I (PH1), idiopathic CaOx stone, enteric hyperoxaluria (EH) and healthy participants) by comparing the number of species and diversity of the microbial populations and pathway for oxalate metabolism by paralleling the gene expression of enzymes involved in oxalate degradation by gut bacteria.

DETAILED DESCRIPTION:
Kidney stones affect as much as 10% of the US population with the most common type of stones made of calcium oxalate. Calcium and oxalate are present in the urine and can bind to each other, and form calcium oxalate kidney stones. Oxalate is absorbed in the gut from the food that is eaten and is removed from the body through urination. Gut bacteria is thought to play a role in decreasing oxalate absorption in the gut and its levels in the urine. With this research we hope to learn about differences in the bacteria that live in the gut of different groups of participants who are likely to form kidney stones, as well as healthy individuals. We will study healthy people with no history of kidney stones, people with a history of calcium oxalate (CaOx) kidney stones, people with a genetic disease called primary hyperoxaluria type1 (PH1) that increases their chances to form calcium oxalate kidney stones and, people with enteric hyperoxaluria (EH) a disease in which individuals have short bowels due to surgery which lead them to get calcium oxalate kidney stones.

Our research questions are:

1. How different is the gut bacteria between participants with the conditions that make them more likely to form kidney stones and healthy participants with no history of kidney stones?
2. Is there any difference in the function of the individual bacteria, Oxalobacter formigenes known to reduce oxalate, between healthy participants with no history kidney stones and participants with PH1?

ELIGIBILITY:
Inclusion Criteria:

* Primary hyperoxaluria: Patients diagnosed with type I PH by genetic testing and part of the Rare Kidney Stone Consortium (RKSC) Primary hyperoxaluria registry
* Enteric hyperoxaluria: Patients with Roux-en-Y-gastric-bypass
* Idiopathic CaOx stone : History of passing or having surgically removed a calcium oxalate kidney stone within 5 years of recruitment
* Healthy participants with no history of kidney or bowel disease

Exclusion Criteria:

* History of kidney or liver transplant
* History of antibiotics use within 6 months of recruitment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a cross sectional study with 60 patients that will collect 2 fecal samples within one week. We will include:
  * 15 participants with healthy kidney function
  * 15 participants with Calcium Oxalate kidney stone(s)
  * 15 participants with Primary Hyperoxaluria type I
  * 15 participants with Enteric Hyperoxaluria
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Differences in composition of the fecal microbiome as measured by 16S ribosomal ribonucleic acid (rRNA) sequencing and whole genome shotgun sequencing between the study groups. | 1 year
  Diversity and abundance of operational taxonomic units (OTUs) between different groups of subjects will be tested. Data from shotgun sequencing and degenerate quantitative polymerase chain reactions (qPCRs) will yield comparative expressions of the oxalate metabolism genes between the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University School of Medicine, New York, New York, United States